CLINICAL TRIAL: NCT04486729
Title: Respiratory System Mechanics and Gas Exchange Characteristics Applying Different Ventilatory Strategies in Patients With SARS-CoV-2
Brief Title: Respiratory Mechanics and Gas Exchange Characteristics in Patient With SARS-CoV-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanatorio Anchorena San Martin (Other)
Responsible Party: Principal Investigator, Matias Accoce, Head of physical therapy department, Sanatorio Anchorena San Martin
Other Study IDs: 10.2020
Record Dates: First submitted 2020-07-21; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Covid19; ARDS, Human
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: High PEEP with end inspiratory pause — Applying a PEEP value 10 cmH2O higher than the lower inflection point of the pressure-volume curve of the respiratory system with end inspiratory pause addition in volumen control ventilation
Other: Low PEEP - FiO2 high — Applying a PEEP value equal to the lower inflection point of the pressure-volume curve of the respiratory system with a FiO2 necessary to achieve a SpO2 96-98%
Other: High PEEP without end inspiratory pause — Applying a PEEP value 10 cmH2O higher than the lower inflection point of the pressure-volume curve of the respiratory system without end inspiratory pause addition in volumen control ventilation
Other: Low PEEP - FiO2 low — Applying a PEEP value equal to the lower inflection point of the pressure-volume curve of the respiratory system with a FiO2 necessary to achieve a SpO2 88-92%

SUMMARY:
The combination of different ventilatory strategies and its effects on respiratory mechanics and gas exchange in patients under mechanical ventilation with acute respiratory distress syndrome secondary to coronavirus-19 has been scarcely described.

DETAILED DESCRIPTION:
Investigation in mechanically ventilated patients with with acute respiratory distress syndrome (ARDS) secondary to coronavirus-19 (COVID-19) is emerging due to presumed differences with typical ARDS from other origin. Considering these issues, the effects of ventilatory strategies such as positive end expiratory pressure, end inspiratory pause and fraction of inspired oxygen on respiratory mechanics and gas exchange must be studied in order to characterize the behavior of COVID-19 ARDS during invasive mechanical ventilation and choose the best combination of ventilatory settings.

In this study the investigators will evaluate the changes in respiratory mechanics and gas exchange produced by low and high positive end expiratory pressure, low and high inspired oxygen fraction and the application of end inspiratory pause during volume controlled mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* less than 72 hs since ARDS diagnosis
* Moderate to severe ARDS
* central venous catheter and arterial line available
* Need of neuromuscular blocking agents
* Supine position
* Informed consent accepted
* Airway opening pressure lower than 20 cmH2O

Exclusion Criteria:

* RASS target higher than -5
* COPD diagnosis
* Pneumothorax
* Intracraneal Hypertension
* Pregnancy
* Cardiac inssuficiency uncompensated
* Chest wall deformity
* Bronchopleural fistula
* Contraindication to use esophageal manometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS secondary to COVID-19 under invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-10 (Estimated); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
Driving transpulmonary pressure (cmH2O) | 10 minutes
  The driving transpulmonary pressure will be evaluated between the high and low PEEP condition using the formula: driving transpulmonary pressure = driving airway pressure - driving esophageal pressure (cmH2O).
Bohr dead space fraction (%) | 10 minutes
  The Bohr dead space fraction will be evaluated with high PEEP between the condition with end inspiratory pause and with no end inspiratory pause application using the formula: Bohr dead space fraction = Alveolar pressure of CO2 (PACO2) - Expired pressure of CO2 (PECO2) / PACO2
Shunt fraction (%) | 10 minutes
  The shunt fraction will be evaluated with low PEEP between the condition with high fraction of oxygen to achieve a saturation goal of 96-98% and the condition with low fraction of oxygen to achieve a saturation goal of 88-92%. The shunt fraction will be calculated using the formula: Qs/Qt = (capillary oxygen content - arterial oxygen content)/(capillary oxygen content - venous oxygen content)

CONTACTS AND LOCATIONS:
Locations (1):
- Sanatorio Anchorena San Martin, San Martín, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Ziehr DR, Alladina J, Petri CR, Maley JH, Moskowitz A, Medoff BD, Hibbert KA, Thompson BT, Hardin CC. Respiratory Pathophysiology of Mechanically Ventilated Patients with COVID-19: A Cohort Study. Am J Respir Crit Care Med. 2020 Jun 15;201(12):1560-1564. doi: 10.1164/rccm.202004-1163LE. No abstract available. PMID 32348678
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Gattinoni L, Chiumello D, Caironi P, Busana M, Romitti F, Brazzi L, Camporota L. COVID-19 pneumonia: different respiratory treatments for different phenotypes? Intensive Care Med. 2020 Jun;46(6):1099-1102. doi: 10.1007/s00134-020-06033-2. Epub 2020 Apr 14. No abstract available. PMID 32291463
- [Background] Chen L, Del Sorbo L, Grieco DL, Junhasavasdikul D, Rittayamai N, Soliman I, Sklar MC, Rauseo M, Ferguson ND, Fan E, Richard JM, Brochard L. Potential for Lung Recruitment Estimated by the Recruitment-to-Inflation Ratio in Acute Respiratory Distress Syndrome. A Clinical Trial. Am J Respir Crit Care Med. 2020 Jan 15;201(2):178-187. doi: 10.1164/rccm.201902-0334OC. PMID 31577153
- [Background] Tusman G, Gogniat E, Madorno M, Otero P, Dianti J, Ceballos IF, Ceballos M, Verdier N, Bohm SH, Rodriguez PO, San Roman E. Effect of PEEP on Dead Space in an Experimental Model of ARDS. Respir Care. 2020 Jan;65(1):11-20. doi: 10.4187/respcare.06843. Epub 2019 Oct 15. PMID 31615922
- [Background] Aguirre-Bermeo H, Moran I, Bottiroli M, Italiano S, Parrilla FJ, Plazolles E, Roche-Campo F, Mancebo J. End-inspiratory pause prolongation in acute respiratory distress syndrome patients: effects on gas exchange and mechanics. Ann Intensive Care. 2016 Dec;6(1):81. doi: 10.1186/s13613-016-0183-z. Epub 2016 Aug 24. PMID 27558174
- [Background] Santos C, Ferrer M, Roca J, Torres A, Hernandez C, Rodriguez-Roisin R. Pulmonary gas exchange response to oxygen breathing in acute lung injury. Am J Respir Crit Care Med. 2000 Jan;161(1):26-31. doi: 10.1164/ajrccm.161.1.9902084. PMID 10619793
- [Background] Pan C, Chen L, Lu C, Zhang W, Xia JA, Sklar MC, Du B, Brochard L, Qiu H. Lung Recruitability in COVID-19-associated Acute Respiratory Distress Syndrome: A Single-Center Observational Study. Am J Respir Crit Care Med. 2020 May 15;201(10):1294-1297. doi: 10.1164/rccm.202003-0527LE. No abstract available. PMID 32200645
- [Background] Chen L, Del Sorbo L, Grieco DL, Shklar O, Junhasavasdikul D, Telias I, Fan E, Brochard L. Airway Closure in Acute Respiratory Distress Syndrome: An Underestimated and Misinterpreted Phenomenon. Am J Respir Crit Care Med. 2018 Jan 1;197(1):132-136. doi: 10.1164/rccm.201702-0388LE. No abstract available. PMID 28557528
- [Background] Tobin MJ. Basing Respiratory Management of COVID-19 on Physiological Principles. Am J Respir Crit Care Med. 2020 Jun 1;201(11):1319-1320. doi: 10.1164/rccm.202004-1076ED. No abstract available. PMID 32281885
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Background] Yoshida T, Amato MBP, Grieco DL, Chen L, Lima CAS, Roldan R, Morais CCA, Gomes S, Costa ELV, Cardoso PFG, Charbonney E, Richard JM, Brochard L, Kavanagh BP. Esophageal Manometry and Regional Transpulmonary Pressure in Lung Injury. Am J Respir Crit Care Med. 2018 Apr 15;197(8):1018-1026. doi: 10.1164/rccm.201709-1806OC. PMID 29323931
- [Background] Tahvanainen J, Meretoja O, Nikki P. Can central venous blood replace mixed venous blood samples? Crit Care Med. 1982 Nov;10(11):758-61. doi: 10.1097/00003246-198211000-00012. PMID 7140317
- [Background] Monnet X, Teboul JL. Passive leg raising: five rules, not a drop of fluid! Crit Care. 2015 Jan 14;19(1):18. doi: 10.1186/s13054-014-0708-5. No abstract available. PMID 25658678
- [Background] Iannuzzi M, De Sio A, De Robertis E, Piazza O, Servillo G, Tufano R. Different patterns of lung recruitment maneuvers in primary acute respiratory distress syndrome: effects on oxygenation and central hemodynamics. Minerva Anestesiol. 2010 Sep;76(9):692-8. Epub 2010 May 14. PMID 20820146
- [Background] Odenstedt H, Lindgren S, Olegard C, Erlandsson K, Lethvall S, Aneman A, Stenqvist O, Lundin S. Slow moderate pressure recruitment maneuver minimizes negative circulatory and lung mechanic side effects: evaluation of recruitment maneuvers using electric impedance tomography. Intensive Care Med. 2005 Dec;31(12):1706-14. doi: 10.1007/s00134-005-2799-6. Epub 2005 Sep 22. PMID 16177920
- [Derived] Dorado JH, Perez J, Navarro E, Gogniat E, Torres S, Cagide S, Accoce M. Impact of liberal versus conservative saturation targets on gas exchange indices in COVID-19 related acute respiratory distress syndrome: a physiological study. Rev Bras Ter Intensiva. 2021 Oct-Dec;33(4):537-543. doi: 10.5935/0103-507X.20210081. Epub 2022 Jan 24. PMID 35081237